CLINICAL TRIAL: NCT06829381
Title: Tailoring One-Anastomosis Gastric Bypass Based on Total Small Bowel Length - A Randomized Controlled Trial
Brief Title: Tailored One Anastomosis Gastric Bypass
Acronym: OAGB-TL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, Shmuel Kivity, MD, Dr Adam-Abu Abeid - Assistant Professor, Consultant Bariatric Surgeon, Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TLV-0586-24
Record Dates: First submitted 2025-02-11; First posted 2025-02-17 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Metabolic and Bariatric Surgery
Keywords: one anastomosis gastric bypass; obesity; weight loss; tailoring
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group BPL 180 cm (Active Comparator): Total bowel length measure and BPL will be 180 cm regardless of total small bowel length
  Interventions: Procedure: Control - BPL 180 cm
- Tailored BPL length (Experimental): Total bowel length measure and BPL will be 40% of total bowel length ensuring at least 250 cm common channel
  Interventions: Procedure: Tailored BPL length

INTERVENTIONS:
Procedure: Tailored BPL length — Total bowel length measure and BPL will be 40% of total bowel length ensuring at least 250 cm common channel
  Arms: Tailored BPL length
Procedure: Control - BPL 180 cm — Total bowel length measure and BPL will be180 cm
  Arms: Control group BPL 180 cm

SUMMARY:
One Anastomosis Gastric Bypass (OAGB) is the most common metabolic and bariatric surgery (MBS) in Israel, recognized for its effectiveness in achieving sustainable weight loss and mitigating obesity-related diseases. The metabolic outcomes of OAGB are significantly influenced by the length of the biliopancreatic limb (BPL). The objective of this study is to determine whether tailoring the BPL length to the total small bowel length (TSBL) results in more effective weight loss compared to patients undergoing OAGB with a fixed BPL of 180 cm. Efficacy and safety of this approach will also be evaluated, ensuring it does not lead to long-term morbidity or negatively impact patients' quality of life.

DETAILED DESCRIPTION:
Scientific Background and Rationale for the Study One-Anastomosis Gastric Bypass (OAGB) is the most common bariatric procedure in Israel [1]. Over the years, OAGB has been proven to be an effective surgery, yielding significant and sustained weight loss, improvement in obesity-related comorbidities, and a relatively low failure rate [2].

The procedure involves separating a long gastric pouch from the remaining stomach and creating an anastomosis between the pouch and a distant loop of the small intestine [3]. Since this procedure bypasses a relatively long intestinal segment (typically 150-200 cm), it results in malabsorption of carbohydrates, fats, proteins, and other nutrients. This malabsorption-related mechanism leads to greater weight loss compared to purely restrictive surgeries like sleeve gastrectomy [4].

The length of the bypassed segment, specifically the biliopancreatic limb (BPL), plays a critical role in determining the metabolic outcomes of OAGB. A longer BPL is associated with more significant weight loss and greater improvement in obesity-related diseases [5]. However, the ideal BPL length remains a topic of global debate. Some experts recommend measuring the total small bowel length (TSBL) or ensuring at least 250-300 cm of common channel (CC) to prevent pathological malabsorption in patients with a shorter bowel and to reduce the risk of weight regain in those with a longer bowel [3,6].

Currently, the most widely accepted approach is to standardize the BPL length at 150-200 cm, as studies have shown that this range minimizes the risk of nutritional deficiencies [7]. However, tailoring the BPL length to the patient's TSBL is an increasingly recognized strategy that may optimize outcomes by ensuring a more precise CC length, thereby reducing complications and improving long-term weight loss.

Study Objective To evaluate whether tailoring the BPL length to the TSBL results in more effective weight loss compared to a standard bypass length of 180 cm.

Study Endpoints BPL and TSBL lengths Weight progression during follow-up Postoperative nutritional complications Improvement in obesity-related comorbidities Study Participants Single-center cohort: 200 patients Multi-center cohort: 500 patients Participating centers: Ichilov Medical Center, Assuta Tel Aviv, Herzliya Medical Center Participant Recruitment and Informed Consent Process

Eligible participants (competent adults) will be invited to sign a digital informed consent form via the PM7 system. The process includes:

A face-to-face explanation Time for consideration An opportunity to ask questions The signed consent form will be stored digitally in PM7 and printed as needed. If digital signing is not possible, a paper form will be used. The process adheres to Regulation 169 and follows an updated consent protocol. Enrollment and consent will take place during the preoperative consultation at the bariatric clinic.

Inclusion Criteria Patients aged 18 and older scheduled for OAGB at Tel Aviv Sourasky Medical Center Exclusion Criteria Special populations - Patients under 18, pregnant women, individuals lacking decision-making capacity, etc.

Previous bariatric surgery Withdrawal Criteria TSBL < 450 cm, as this would prevent achieving a common channel length of at least 250-300 cm, increasing the risk of severe malabsorption and nutritional deficiencies (protein, vitamins, iron).

Study Methods and Design Randomization Process After enrollment and consent, participants will be randomly assigned to either the intervention or control group.

Surgical Interventions Intervention Group: The surgeon will manually measure TSBL intraoperatively and create a BPL equal to 40% of the TSBL. This ensures a minimum CC length of 250-300 cm, in line with standard OAGB recommendations.

Control Group: The surgeon will measure the TSBL but will create a fixed BPL of 180 cm, as per the current standard.

Postoperative Follow-Up Patients will undergo routine follow-up at 2 weeks, 1, 3, 6, and 12 months, and annually thereafter.

Data Collection and Privacy Identifiable patient information will be separated from the dataset by an authorized investigator.

The principal investigator will maintain the coding key in a password-protected file within the hospital network.

Data will remain within the hospital and not be shared externally. Statistical Analysis T-tests and chi-square tests will be used to compare baseline characteristics. Results will be reported in tables with standard deviation and p-values. Study Timeline and Duration Total study duration: 8 years from approval.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years) undergoing OAGB

Exclusion Criteria:

* Patients <18 years, pregnant women, or those lacking decision-making capacity Prior bariatric surgery Short bowel (<450 cm)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-01-29 (Actual); Primary Completion 2029-01-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
weight loss | 6 months, one year, and 3 years after surgery
  Total weight loss will be calculated as - preoperative weight-last follow-up weight/preoperative weight * 100

SECONDARY OUTCOMES:
Postoperative nutritional complications | 6 months and one year after surgery
  Postoperative nutritional complications - albumin, vitamins, iron
resolution of obesity related diseases | 6 months and one year postopertively
  Resolution of obesity related diseases - Type 2 diabetes, hypertension, hyperlipidemia.
  Resolution of diseases definition - If patients no longer required medications or other treatment methods prior to surgery. In case of type 2 diabetes, a value of Hba1c below 6.5% in addition to cessation of antidiabetic to define its resolution.
Bariatric Analysis and Reporting Outcome System score | 6 months and one year postopertively
  Bariatric Analysis and Reporting Outcome System score - quality of life assessment.
  The assessment will be as follows - ≥7.0 - Excellent 5.1 - 6.9 - Very Good 3.1 - 5.0 - Good 1.1 - 3.0 - Fair
  ≤1.0 - Failure Maximum score - 9 (in case of optimal condition and no complications occur) Minimum scire - Negative values (if severe complications occur).
Fecal Score | 6 months, 1 year and 3 years
  Altered bowel habits-such as loose stools, increased frequency of defecation, and even fecal incontinence-can significantly impact quality of life following bariatric surgery. To evaluate these changes, we are using the semi-quantitative Stool Frequency and Consistency Score, also known as the Fecal Score (FS), to assess bowel movement patterns at 6, 12, and 36 months postoperatively. The FS (Fecal Score) is calculated based on fecal frequency and consistency. Fecal frequency is assessed using a 5-point scale: less than twice per week (1 point), every two days (2 points), once daily (3 points), twice daily (4 points), and more than twice daily (5 points). Fecal consistency is also scored on a 5-point scale: watery stools (5 points), loose stools (4 points), normal stools (3 points), firm stools (2 points), and hard stools associated with constipation (1 point). The FS is derived by summing the fecal frequency and consistency scores.

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Slagter N, de Heide LJM, Jutte EH, Kaijser MA, Damen SL, van Beek AP, Emous M. Tailoring limb length based on total small bowel length in one anastomosis gastric bypass surgery (TAILOR study): study protocol for a randomized controlled trial. Trials. 2022 Jun 22;23(1):526. doi: 10.1186/s13063-022-06456-w. PMID 35733198
- [Background] Hany M, Zidan A, Aboelsoud MR, Torensma B. Laparoscopic sleeve gastrectomy vs one-anastomosis gastric bypass 5-year follow-up: a single-blinded randomized controlled trial. J Gastrointest Surg. 2024 May;28(5):621-633. doi: 10.1016/j.gassur.2024.01.038. Epub 2024 Feb 9. PMID 38704199
- [Background] Kansou G, Lechaux D, Delarue J, Badic B, Le Gall M, Guillerm S, Bail JP, Thereaux J. Laparoscopic sleeve gastrectomy versus laparoscopic mini gastric bypass: One year outcomes. Int J Surg. 2016 Sep;33 Pt A:18-22. doi: 10.1016/j.ijsu.2016.07.051. Epub 2016 Jul 22. PMID 27452299
- [Background] Jones NR, McCormack T, Constanti M, McManus RJ. Diagnosis and management of hypertension in adults: NICE guideline update 2019. Br J Gen Pract. 2020 Jan 30;70(691):90-91. doi: 10.3399/bjgp20X708053. Print 2020 Feb. No abstract available. PMID 32001477
- [Background] Riddle MC, Cefalu WT, Evans PH, Gerstein HC, Nauck MA, Oh WK, Rothberg AE, le Roux CW, Rubino F, Schauer P, Taylor R, Twenefour D. Consensus Report: Definition and Interpretation of Remission in Type 2 Diabetes. Diabetes Care. 2021 Aug 30;44(10):2438-44. doi: 10.2337/dci21-0034. Online ahead of print. PMID 34462270
- [Background] Schijns W, Aarts EO, Berends FJ, Janssen IM, Schweitzer DH. Loose and frequent stools and PTH levels are positively correlated post-gastric bypass surgery due to less efficient intestinal calcium absorption. Surg Obes Relat Dis. 2016 Sep-Oct;12(8):1548-1553. doi: 10.1016/j.soard.2016.04.011. Epub 2016 Apr 13. PMID 27396549
- [Background] Oria HE, Moorehead MK. Updated Bariatric Analysis and Reporting Outcome System (BAROS). Surg Obes Relat Dis. 2009 Jan-Feb;5(1):60-6. doi: 10.1016/j.soard.2008.10.004. Epub 2008 Nov 1. PMID 19161935
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Abu-Abeid A, Vitiello A, Berardi G, Dayan D, Velotti N, Schiavone V, Franzese A, Musella M. Implementation of updated enhanced recovery after bariatric surgery guidelines: adapted protocol in a single tertiary center. Updates Surg. 2024 Aug;76(4):1397-1404. doi: 10.1007/s13304-024-01824-4. Epub 2024 Mar 28. PMID 38546967
- [Background] Felsenreich DM, Langer FB, Eichelter J, Jedamzik J, Gensthaler L, Nixdorf L, Gachabayov M, Rojas A, Vock N, Zach ML, Prager G. Bariatric Surgery-How Much Malabsorption Do We Need?-A Review of Various Limb Lengths in Different Gastric Bypass Procedures. J Clin Med. 2021 Feb 10;10(4):674. doi: 10.3390/jcm10040674. PMID 33578635
- [Background] Butler AA, O'Rourke RW. Bariatric surgery in the era of personalized medicine. Gastroenterology. 2013 Mar;144(3):497-500. doi: 10.1053/j.gastro.2013.01.027. Epub 2013 Jan 21. No abstract available. PMID 23347671
- [Background] Thanos PK, Hanna C, Mihalkovic A, Hoffman AB, Posner AR, Busch J, Smith C, Badgaiyan RD, Blum K, Baron D, Mastrandrea LD, Quattrin T. The First Exploratory Personalized Medicine Approach to Improve Bariatric Surgery Outcomes Utilizing Psychosocial and Genetic Risk Assessments: Encouraging Clinical Research. J Pers Med. 2023 Jul 20;13(7):1164. doi: 10.3390/jpm13071164. PMID 37511777
- [Background] Soong TC, Almalki OM, Lee WJ, Ser KH, Chen JC, Wu CC, Chen SC. Measuring the small bowel length may decrease the incidence of malnutrition after laparoscopic one-anastomosis gastric bypass with tailored bypass limb. Surg Obes Relat Dis. 2019 Oct;15(10):1712-1718. doi: 10.1016/j.soard.2019.08.010. Epub 2019 Aug 21. PMID 31558409
- [Background] Abu-Abeid A, Bendayan A, Yuval JB, Eldar SM, Lahat G, Lessing Y. Primary versus Revisional One Anastomosis Gastric Bypass: Outcomes of Patients with at Least 8-Year Follow-Up. Obes Facts. 2024;17(3):303-310. doi: 10.1159/000538768. Epub 2024 Apr 9. PMID 38593760
- [Background] Shahmiri SS, Pazouki A, Jazi AHD, Safari S, Mahjoubi M, Sheikhbahaei E, Kermansaravi M. Long-Term Weight Loss Outcomes of One Anastomosis Gastric Bypass: Assessment of 1971 Patients with 5-9-Year Follow-Up. Obes Surg. 2025 Jan;35(1):102-111. doi: 10.1007/s11695-024-07618-2. Epub 2024 Dec 14. PMID 39674852
- [Background] Angrisani L, Santonicola A, Iovino P, Palma R, Kow L, Prager G, Ramos A, Shikora S; Collaborative Study Group for the IFSO Worldwide Survey. IFSO Worldwide Survey 2020-2021: Current Trends for Bariatric and Metabolic Procedures. Obes Surg. 2024 Apr;34(4):1075-1085. doi: 10.1007/s11695-024-07118-3. Epub 2024 Mar 4. PMID 38438667
- [Background] Bekheit M, Ibrahim MY, Tobar W, Galal I, Elward AS. Correlation Between the Total Small Bowel Length and Anthropometric Measures in Living Humans: Cross-Sectional Study. Obes Surg. 2020 Feb;30(2):681-686. doi: 10.1007/s11695-019-04238-z. PMID 31686382
- [Background] Pizza F, D'Antonio D, Lucido FS, Tolone S, Dell'Isola C, Gambardella C. Postoperative Clinical-Endoscopic Follow-up for GERD and Gastritis After One Anastomosis Gastric Bypass for Morbid Obesity: How, When, and Why. Obes Surg. 2020 Nov;30(11):4391-4400. doi: 10.1007/s11695-020-04805-9. Epub 2020 Jul 3. PMID 32621053
- [Background] Carbajo MA, Luque-de-Leon E, Jimenez JM, Ortiz-de-Solorzano J, Perez-Miranda M, Castro-Alija MJ. Laparoscopic One-Anastomosis Gastric Bypass: Technique, Results, and Long-Term Follow-Up in 1200 Patients. Obes Surg. 2017 May;27(5):1153-1167. doi: 10.1007/s11695-016-2428-1. PMID 27783366
- [Background] Almuhanna M, Soong TC, Lee WJ, Chen JC, Wu CC, Lee YC. Twenty years' experience of laparoscopic 1-anastomosis gastric bypass: surgical risk and long-term results. Surg Obes Relat Dis. 2021 May;17(5):968-975. doi: 10.1016/j.soard.2021.01.010. Epub 2021 Jan 21. PMID 33619007
- [Derived] Abu-Abeid A, Ovadya R, Gosher N, Yuval JB, Bendayan A, Keidar A, Eldar SM. Tailored Biliopancreatic Limb Length to 40% of Total Small Bowel Length in One Anastomosis Gastric Bypass (TABLE-40): Protocol of a Prospective Randomized Controlled Trial. Obes Surg. 2025 Sep;35(9):3619-3625. doi: 10.1007/s11695-025-08035-9. Epub 2025 Jul 10. PMID 40638030